CLINICAL TRIAL: NCT04045600
Title: Stimulus Control Refinements of Functional Communication Training
Brief Title: Refinements of Functional Communication Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Wayne W. Fisher, Ph.D., BCBA-D, LP, Henry Rutgers Endowed Professor of Pediatrics, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro2019001493
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Aggression; Self-injurious Behavior
MeSH Terms: conditions — Aggression; Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mult FCT/Trad FCT (Experimental): Participants assigned to this condition will receive both traditional FCT (trad FCT) and FCT with multiple schedules (mult FCT) to evaluate the effects of mult FCT on renewal, super-resurgence, and reinstatement.
  Interventions: Behavioral: Trad FCT; Behavioral: Mult FCT
- Mult FCT + Stimulus Fading/Trad FCT (Experimental): Participants assigned to this condition will receive both traditional FCT (trad FCT) and FCT with multiple schedules and stimulus fading (mult FCT + stimulus fading) to evaluate the effects of mult FCT and gradual fading of contextual stimuli on renewal, super-resurgence, and reinstatement.
  Interventions: Behavioral: Trad FCT; Behavioral: Mult FCT + Stimulus Fading

INTERVENTIONS:
Behavioral: Trad FCT — This intervention emulates a traditional reinforcement schedule-thinning method during FCT in which clinicians program delays to reinforcement without discriminative stimuli (e.g., the child learns that some FCRs result in reinforcement and some do not). By programming reinforcement approximately every 15 s, the rate of reinforcement will be equivalent to mult FCT. During Period 1 of this project, trad FCT served as an appropriate control condition to which mult FCT could be compared.
Behavioral: Mult FCT — This intervention involves correlating discriminative stimuli (e.g., purple and yellow index cards) with times in which reinforcement for the functional communication response (FCR) is and is not available. During Period 1 of this project, this procedure resulted in rapid reduction of destructive behavior and mitigated resurgence and renewal when the discriminative stimuli were used as programmed.
  Arms: Mult FCT/Trad FCT
Behavioral: Mult FCT + Stimulus Fading — This condition is similar to mult FCT except that the experimenters will gradually incorporate natural stimuli (e.g., rugs, tables, lamps) into sessions to approximate target settings that may occasion relapse typically without such gradual stimulus fading.
  Arms: Mult FCT + Stimulus Fading/Trad FCT

SUMMARY:
Although treatments for problem behavior, like functional communication training (FCT), can be highly effective in the clinic, changes in the way the FCT is implemented (e.g., when transferring treatment to the home, when teachers implement treatment with poor fidelity) can result in treatment relapse. The goal of this study is to evaluate whether using treatment signals and gradually introducing materials from natural contexts can help mitigate treatment relapse during context changes and poor treatment-integrity scenarios.

DETAILED DESCRIPTION:
The most common treatment for problem behavior is functional communication training (FCT). FCT involves teaching children to request what they want, rather than engaging in problem behavior when they don't get their way, and then teach them that they cannot always ask for their way and instead must wait or work appropriately first. While FCT is effective, problem behavior sometimes comes back after treatment when children encounter treatment challenges, like long periods of not getting their way, when caregivers deliver treatment differently than what they are used to (e.g., caregivers delivering FCT incorrectly), or experiencing treatment in a new place (e.g., the home, the classroom). The purpose of this research study is to determine whether the experimenters can reduce the chances of children returning to problem behavior during these challenges by teaching them to pay attention to treatment signals (e.g., a red card that indicates treatment is in place) and gradually changing the treatment setting to appear more like the home or classroom. First, the experimenters will provide each child with their way in a home-like environment containing a couch, rug, etc. Next, within a barren therapy room, the experimenters will conduct two of the following three types of treatments: (1) a treatment with no signals that indicate when their child can and cannot have their way, (2) a treatment with signals, and (3) a treatment with signals plus introduction of items from the natural environment such as rugs and couches. Then, the experimenters will introduce three common treatment challenges in a row to determine whether treatment signals reduce relapse of problem behavior. First, the experimenters will introduce the treatments in the home-like environment to see if the child continues to respond appropriately in a setting different than the therapy room. Second, the experimenters will simulate a transition to the school by having the child experience treatment in a classroom-like environment (e.g., with desks and chalkboards) while the teacher makes the child wait a long period of time to get their way. This would be similar to when a teacher cannot give the child attention or a preferred item because they are busy with other students. Third, the experimenters will simulate the teacher implementing treatment differently than the child is used to in the classroom by the teacher delivering preferred activities according to a timed schedule rather than when the child asks. This simulates the common event of a teacher delivering preferred activities like breaks or recess regardless of the child's behavior. The goal is to determine how well the treatments perform across each of these common challenges.

ELIGIBILITY:
Inclusion Criteria:

* Boys and girls from ages 3 to 17
* Destructive behavior that occurs at least 10 times a day despite previous treatment
* Destructive behavior reinforced by social consequences like attention (FCT is not appropriate for automatically reinforced destructive behavior)
* On a stable psychoactive drug regimen for at least 10 half-lives per drug or drug free
* Stable educational plan and placement with no anticipated changes during the child's treatment

Exclusion Criteria:

* Patients who do not meet the inclusion criteria
* Patients currently receiving 15 or more hours per week of treatment for their destructive behavior
* DSM-5 diagnosis of Rett syndrome or other degenerative conditions (e.g., inborn error of metabolism)
* A comorbid health condition or major mental disorder that would interfere with study participation
* Occurrence of SIB during study assessments that presents a risk of serious or permanent harm (e.g., detached retinas) based on our routine clinical-risk assessment
* Patients requiring drug-treatment changes, but the experimenters will invite these patients to participate if they meet inclusion criteria after drug regimen is stable.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Destructive Behavior in Renewal Test | Through study completion, an average of 3 weeks.
  The investigators will measure the rate of destructive behavior following successful treatment when the FCT is implemented in a context not associated with treatment (e.g., the baseline, home-like context).
Rate of Destructive Behavior in Super-Resurgence Test | Through study completion, an average of 3 weeks.
  The investigators will measure the rate of destructive behavior when FCT is implemented in a context not associated with treatment (e.g., a classroom context) by an implementer who fails to reinforce the communication response. This would be similar to a busy teacher in a classroom who is unable to attend to the child due to assisting another student.
Rate of Destructive Behavior in Reinstatement Test | Through study completion, an average of 3 weeks.
  The investigators will measure the rate of destructive behavior when FCT is not implemented as prescribed (i.e., reinforcement is delivered on a time-based schedule, rather than following communication responses). This would be similar to a teacher who delivers breaks from work based on the school schedule (e.g., switching from math to reading) rather than the child's request for a break during the math period).

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Fisher, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Children's Specialized Hospital - Rutgers University Center for Autism Research, Education, and Services, Somerset, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
The experimenters plan to make data available to participants, if requested, and submit results for publication.
Supporting Information: Study Protocol, ICF
Time Frame: The informed consent form shall be available to the caregiver immediately after caregiver signature. If requested, the study protocol will be sent to the caregiver after the study is complete.
Access Criteria: Each caregiver of a child enrolled in the study will be eligible to receive the above documents.